CLINICAL TRIAL: NCT01205230
Title: An Open-Label Study to Evaluate the Effects of Ketoconazole and the Effects of Esomeprazole on the Pharmacokinetics of Orally Administered Repeat Doses of Pazopanib in Subjects With Solid Tumor Malignancies
Brief Title: VEG113971: An Open-Label Study of the Effects of Ketoconazole or Esomeprazole on Pazopanib PK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 113971
Record Dates: First submitted 2010-08-12; First posted 2010-09-20 (Estimated); Results first posted 2012-04-24 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Cancer
Keywords: Esomeprazole; Pharmacogenetics; Pharmacokinetics; Ketoconazole; Pazopanib; Drug Interaction; Safety; Solid Tumors
MeSH Terms: conditions — Neoplasms | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pazonib+ketoconazole (Experimental): Administration of oral pazopanib 400mg (2 200-mg tablets) once-daily each morning for at least 7 consecutive doses during Period 1. Then administration of oral ketoconazole 400 mg (2 - 200 mg tablets) followed immediately by pazopanib 400 mg (2 -200 mg tablets) once-daily each morning for a total of 5 consecutive doses during Period 2.
  Interventions: Drug: pazopanib
- Pazonib+esomeprazole (Experimental): Subjects will receive orally administered pazopanib 800mg (4 - 200mg tablets) once-daily each morning for at least 7 consecutive doses in Period 1. In the evening on the last day of Period 1, subjects will take their initial dose of esomeprazole 40 mg (1 - 40 mg capsule) approximately 3 hours after the evening meal. Subjects will continue to receive pazopanib (each morning) and esomeprazole each evening once-daily for a total of 5 consecutive doses.
  Interventions: Drug: pazopanib

INTERVENTIONS:
Drug: pazopanib — Adenosine triphosphate (ATP)-competitive tyrosine kinase inhibitor of vascular endothelial growth factor receptor (VEGFR)-1, -2, and -3, platelet derivative growth factor receptor (PDGFR)
  Other Names: Votrient

SUMMARY:
The purpose of this study is to determine how dosing with ketoconazole (Nizoral) or esomeprazole (Nexium) affects the pharmacokinetics of oral pazopanib. The study will also test for safety of pazopanib when administered with ketoconazole or esomeprazole.

DETAILED DESCRIPTION:
The study is a 2-arm, open-label, repeat-dose, single sequence, crossover, study designed to evaluate the effects of ketoconazole (Arm A) and esomeprazole (Arm B) on the pharmacokinetics (PK) of oral pazopanib in subjects with solid tumor malignancies. This study will compare the PK parameters of oral pazopanib and its metabolite concentrations when given alone and when co-administered with either ketoconazole (Arm A) or esomeprazole (Arm B). Safety assessments (physical examinations, vital signs, 12-lead electrocardiograms, Eastern Cooperative Oncology Group performance status, clinical laboratory assessments, and monitoring of adverse events) will also be evaluated during the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed, written informed consent
* 18 years of age or legal age of consent if greater than 18 years at the time of signing consent
* Histologically confirmed diagnosis of refractory or relapsed advanced solid tumor malignancy after standard therapy OR for which there is no standard therapy OR for which subject opts not to receive standard therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate baseline organ function
* Subjects may not have had a transfusion within 7 days of screening assessment.
* Subjects receiving anticoagulant therapy are eligible if their INR is stable and within the protocol recommended range.
* Male OR
* Female of non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who has had: a hysterectomy, a bilateral oophorectomy (ovariectomy), a bilateral tubal ligation, or is post-menopausal OR
* Non-pregnant Female of childbearing potential, including any female who has had a negative serum pregnancy test within 14 days prior to the first dose of study treatment, agrees to use acceptable contraceptive methods, used consistently and in accordance with both the product label and the instructions of the study physician. OR
* Female, if lactating, agrees to stop nursing prior to first dose until 14 days after last dose of study drug
* Able to swallow and retain orally administered medication

Exclusion Criteria:

* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for 2 months prior to first dose of study drug
* Clinically significant GI abnormalities that may increase the risk for GI bleeding including, but not limited to: active peptic ulcer disease, known intraluminal metastatic lesion/s with risk of bleeding inflammatory bowel disease (e.g., ulcerative colitis, Crohn's disease), or other GI conditions with increased risk of perforation, history of abdominal fistula, GI perforation, or intra abdominal abscess within 28 days prior to beginning study treatment.
* Clinically significant GI abnormalities that may affect absorption of investigational product including, but not limited to: malabsorption syndrome, major resection of the stomach or small bowel.
* Presence of uncontrolled infection.
* Corrected QT interval (QTc) >480 msec.
* History of any one or more of the following cardiovascular conditions within the past 6 months:

cardiac angioplasty or stenting, myocardial infarction,unstable angina,coronary artery bypass graft surgery, symptomatic peripheral vascular disease, Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA).

* Poorly controlled hypertension Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry.
* History of cerebrovascular accident including transient ischemic attack, pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months. Note: Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible.
* Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major).
* Evidence of active bleeding or bleeding diathesis.
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels.
* Hemoptysis in excess of 2.5 mL (or one-half teaspoon) within 8 weeks of first dose of study drug.
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
* Treatment with any of the following anti-cancer therapies: radiation therapy, surgery or tumor embolization within 14 days prior to the first dose of pazopanib OR chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days or 5 half-lives of a drug (whichever is longer) prior to the first dose of pazopanib.
* Any ongoing toxicity from prior anti-cancer therapy that is > Grade 1 (graded by NCI-CTCAE, version 4.0), at the time of enrollment and/or that is progressing in severity, except alopecia as well as stable (>4 weeks) ≤Grade 2 neuropathy or rash.

-Unable or unwilling to discontinue use of protocol-prohibited medications for at least 14 days or 5 half- lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study.

-Use of HRT prior to study enrollment due to the potential for inhibition of cytochrome P450 enzymes that metabolize estrogens and progestins (Arm A female subjects only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, New Brunswick, New Jersey
  - GSK Investigational Site, Greenville, South Carolina

REFERENCES:
- [Derived] Tan AR, Gibbon DG, Stein MN, Lindquist D, Edenfield JW, Martin JC, Gregory C, Suttle AB, Tada H, Botbyl J, Stephenson JJ. Effects of ketoconazole and esomeprazole on the pharmacokinetics of pazopanib in patients with solid tumors. Cancer Chemother Pharmacol. 2013 Jun;71(6):1635-43. doi: 10.1007/s00280-013-2164-3. Epub 2013 May 1. PMID 23636448

RESULTS

PARTICIPANT FLOW:
Groups:
- Pazopanib, Followed by Pazopanib + Ketoconazole: Pazopanib 400 milligrams (mg) (2x200 mg tablets) once daily (QD), for at least 7 consecutive days in the morning during Period 1, followed by ketoconazole 400 mg (2x200 mg tablets) QD in combination with pazopanib 400 mg (2x200 mg tablets) QD for 5 consecutive days in the morning during Period 2
- Pazopanib, Followed by Pazopanib + Esomeprazole: Pazopanib 800 mg (4x200 mg tablets) QD, for at least 7 consecutive days in the morning during Period 1, followed by pazopanib 800 mg (4x200 mg tablets) QD in the morning in combination with esomeprazole 40 mg (1x40 mg capsule) QD in the evening (approximately 3 hours after the evening meal) for 5 consecutive days during Period 2
Period: Overall Study
Arm/Group | Pazopanib, Followed by Pazopanib + Ketoconazole | Pazopanib, Followed by Pazopanib + Esomeprazole
Started | 21 | 13
Combination Therapy | 21 | 13
Completed | 16 | 13
Not Completed | 5 | 0
Not completed — Adverse Event | 4 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pazopanib, Followed by Pazopanib + Ketoconazole | Pazopanib, Followed by Pazopanib + Esomeprazole | Total
Number analyzed (Participants) | 21 | 13 | 34
Age Continuous [Mean (Standard Deviation); unit: Years]
  Years | 60.0 (12.27) | 57.9 (13.09) | 59.2 (12.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 10 | 2 | 12
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 1 | 2 | 3
  Asian - Central/South Asian Heritage | 2 | 0 | 2
  Asian - South East Asian Heritage | 1 | 0 | 1
  White - White/Caucasian/European Heritage | 17 | 10 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Plasma Pazopanib Area Under the Concentration-time Curve From Zero (Pre-dose) to 24 Hours (AUC[0-24]) of Pazopanib Alone and of Pazopanib in Combination With Ketoconazole and Esomeprazole
Description: Blood samples for pharmacokinetic (PK) analysis of pazopanib were obtained at pre-dose (within 60 minutes prior to pazopanib administration) and at 1, 2, 3, 4, 6, 8, and 24 hours after pazopanib administration. From the plasma concentration-time curve, the PK parameter AUC(0-24) was determined by standard non-compartmental analysis using WinNonlin. Plasma AUC(0-24) is a measure of the amount of drug a participant has been exposed to in 24 hours.
Time Frame: Day 7 of Period 1 (monotherapy) and Day 5 (Study Day 12) of Period 2 (combination therapy). Blood samples were obtained within 60 minutes prior to pazopanib administration and at 1, 2, 3, 4, 6, 8, and 24 hours after pazopanib administration.
Population: Pharmacokinetic (PK) Population: all participants who underwent plasma PK sampling and had evaluable PK assay results from at least one analyte
Measure: Geometric Mean (95% Confidence Interval); unit: Hour*micrograms/milliliters (hr*mcg/mL)
Groups:
- Pazopanib 400 mg QD: Pazopanib 400 milligrams (mg) (2x200 mg tablets) once daily (QD), for at least 7 consecutive days in the morning during Period 1
- Pazopanib 400 mg QD + Ketoconazole 400 mg QD: Ketoconazole 400 mg (2x200 mg tablets) QD in combination with pazopanib 400 mg (2x200 mg tablets) QD for 5 consecutive days in the morning during Period 2
- Pazopanib 800 mg QD: Pazopanib 800 mg (4x200 mg tablets) QD, for at least 7 consecutive days in the morning during Period 1
- Pazopanib 800 mg QD + Esomeprazole 40 mg QD: Pazopanib 800 mg (4x200 mg tablets) QD in the morning in combination with esomeprazole 40 mg (1x40 mg capsule) QD in the evening (administered 1 hour after the evening meal) for 5 consecutive days during Period 2
Arm/Group | Pazopanib 400 mg QD | Pazopanib 400 mg QD + Ketoconazole 400 mg QD | Pazopanib 800 mg QD | Pazopanib 800 mg QD + Esomeprazole 40 mg QD
Number analyzed (Participants) | 21 | 16 | 12 | 12
Hour*micrograms/milliliters (hr*mcg/mL) | 786 [632 to 976] | 1300 [1030 to 1620] | 848 [660 to 1090] | 512 [418 to 627]
Statistical Analysis 1: Comparison: Pazopanib 400 mg QD vs Pazopanib 400 mg QD + Ketoconazole 400 mg QD; Test type: Superiority or Other; Ratio of least square geometric means = 1.66, 90% CI 2-sided [1.39 to 1.99] — Ratio of least square (LS) geometric means (Pazopanib + Ketoconozole : Pazopanib alone)
Statistical Analysis 2: Comparison: Pazopanib 800 mg QD vs Pazopanib 800 mg QD + Esomeprazole 40 mg QD; Test type: Superiority or Other; Ratio of LS geometric means = 0.60, 90% CI 2-sided [0.52 to 0.70] — Ratio of LS geometric means (Pazopanib + Esomeprazole : Pazopanib alone)

2. Primary Outcome: Plasma Maximum Observed Concentration (Cmax) of Pazopanib Alone and of Pazopanib in Combination With Ketoconazole and Esomeprazole
Description: Blood samples for PK analysis of pazopanib were obtained at pre-dose (within 60 minutes prior to pazopanib administration) and at 1, 2, 3, 4, 6, 8, and 24 hours after pazopanib administration. From the plasma concentration-time curve, the PK parameter Cmax was determined by standard non-compartmental analysis using WinNonlin. The concentration-time curve is the result of time points of blood sampling and its measured concentration of pazopanib in the plasma.
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | Pazopanib 400 mg QD | Pazopanib 400 mg QD + Ketoconazole 400 mg QD | Pazopanib 800 mg QD | Pazopanib 800 mg QD + Esomeprazole 40 mg QD
Number analyzed (Participants) | 21 | 16 | 12 | 12
mcg/mL | 40.7 [32.8 to 50.6] | 59.2 [45.1 to 77.6] | 48.9 [39.5 to 60.6] | 28.4 [23.8 to 33.9]
Statistical Analysis 1: Comparison: Pazopanib 400 mg QD vs Pazopanib 400 mg QD + Ketoconazole 400 mg QD; Test type: Superiority or Other; Ratio of LS geometric means = 1.45, 90% CI 2-sided [1.14 to 1.86] — Ratio of LS geometric means (Pazopanib + Ketoconozole : Pazopanib alone)
Statistical Analysis 2: Comparison: Pazopanib 800 mg QD vs Pazopanib 800 mg QD + Esomeprazole 40 mg QD; Test type: Superiority or Other; Ratio of LS geometric means = 0.58, 90% CI 2-sided [0.50 to 0.67] — Ratio of LS geometric means (Pazopanib + Esomeprazole : Pazopanib alone)

3. Primary Outcome: Time of Occurrence of Cmax (Tmax) of Pazopanib Alone and of Pazopanib in Combination With Ketoconazole and Esomeprazole
Description: Blood samples for PK analysis of pazopanib were obtained at pre-dose (within 60 minutes prior to pazopanib administration) and at 1, 2, 3, 4, 6, 8, and 24 hours after pazopanib administration. From the plasma concentration-time curve, the PK parameter tmax was determined by standard non-compartmental analysis using WinNonlin. Nominal data collection time points (TPs) were defined in the protocol; however, the actual data collection TP often differed slightly from the nominal TP for various reasons. This leads to medians and ranges that don't coincide with planned nominal data collection TPs.
Time Frame: as for outcome 1
Population: PK Population
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | Pazopanib 400 mg QD | Pazopanib 400 mg QD + Ketoconazole 400 mg QD | Pazopanib 800 mg QD | Pazopanib 800 mg QD + Esomeprazole 40 mg QD
Number analyzed (Participants) | 21 | 16 | 12 | 12
hours (hr) | 3.48 [2.0 to 24.0] | 3.48 [2.0 to 23.9] | 3 [1.9 to 7.8] | 3.9 [1.0 to 24.8]
Statistical Analysis 1: Comparison: Pazopanib 400 mg QD; Test type: Superiority or Other; Median Difference (Final Values) = -0.45, 90% CI 2-sided [-1.06 to 0.06]
Statistical Analysis 2: Comparison: Pazopanib 800 mg QD vs Pazopanib 800 mg QD + Esomeprazole 40 mg QD; Test type: Superiority or Other; Mean Difference (Final Values) = 1.07, 90% CI 2-sided [-0.10 to 2.44]

4. Secondary Outcome: Plasma Concentration at 24 Hours After Administration (C24) of Pazopanib Alone and of Pazopanib in Combination With Ketoconazole and Esomeprazole
Description: Pazopanib plasma concentration-time data were analyzed by non-compartmental methods with WinNonlin. Calculations were based on the actual sampling times. From the plasma concentration-time data, the PK parameter C24 was determined.
Time Frame: Day 7 of Period 1 (monotherapy) and Day 5 (Study Day 12) of Period 2 (combination therapy). Blood samples were obtained 24 hours after administration of pazopanib.
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | Pazopanib 400 mg QD | Pazopanib 400 mg QD + Ketoconazole 400 mg QD | Pazopanib 800 mg QD | Pazopanib 800 mg QD + Esomeprazole 40 mg QD
Number analyzed (Participants) | 21 | 16 | 12 | 12
mcg/mL | 26.9 [21.5 to 33.6] | 48.7 [36.5 to 65.0] | 27.2 [20.4 to 36.4] | 17.3 [12.6 to 23.7]

5. Secondary Outcome: Plasma AUC(0-24) for the Indicated Metabolites of Pazopanib When Administered Alone or in Combination With Ketoconazole and Ezomeprazole
Description: Blood samples for PK analysis of the metabolites of pazopanib were obtained at pre-dose (within 60 minutes prior to pazopanib administration) and at 1, 2, 3, 4, 6, 8, and 24 hours after pazopanib administration. From the plasma concentration-time curve, the PK parameter AUC(0-24) was determined by standard non-compartmental analysis using WinNonlin. Plasma AUC(0-24) is a measure of the amount of drug a participant has been exposed to in 24 hours.
Time Frame: as for outcome 1
Population: PK Population. One participant from the Pazopanib + Ketoconazole treatment arm was not analyzed for GSK1071306 due to mishandling of PK samples during shipping. Only those participants providing samples were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: hr*mcg/mL
Arm/Group | Pazopanib 400 mg QD | Pazopanib 400 mg QD + Ketoconazole 400 mg QD | Pazopanib 800 mg QD | Pazopanib 800 mg QD + Esomeprazole 40 mg QD
Number analyzed (Participants) | 21 | 16 | 12 | 12
hr*mcg/mL
  GSK1268992, n=21, 16, 12, 12 | 30.3 [23.4 to 39.2] | 30.3 [22.5 to 40.8] | 35.5 [25.4 to 49.6] | 20.8 [16.2 to 26.5]
  GSK1268997, n=20, 13, 12, 12 | 17.4 [13.4 to 22.7] | 6.67 [4.97 to 8.94] | 21.6 [14.2 to 33.0] | 11.2 [7.54 to 16.7]
  GSK1071306, n=21, 15, 12, 12 | 7.61 [5.81 to 9.97] | 4.26 [3.44 to 5.27] | 11.7 [8.24 to 16.6] | 8.14 [5.73 to 11.6]

6. Secondary Outcome: Plasma Cmax for the Indicated Metabolites of Pazopanib When Administered Alone or in Combination With Ketoconazole and Ezomeprazole
Description: Blood samples for PK analysis of the metabolites of pazopanib were obtained at pre-dose (within 60 minutes prior to pazopanib administration) and at 1, 2, 3, 4, 6, 8, and 24 hours after pazopanib administration. From the plasma concentration-time curve, the PK parameter Cmax was determined by standard non-compartmental analysis using WinNonlin. The concentration-time curve is the result of time points of blood sampling and its measured concentration of pazopanib in the plasma.
Time Frame: as for outcome 1
Population: PK Population
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | Pazopanib 400 mg QD | Pazopanib 400 mg QD + Ketoconazole 400 mg QD | Pazopanib 800 mg QD | Pazopanib 800 mg QD + Esomeprazole 40 mg QD
Number analyzed (Participants) | 21 | 16 | 12 | 12
mcg/mL
  GSK1268992 | 1.55 [1.19 to 2.03] | 1.52 [1.16 to 2.01] | 1.95 [1.48 to 2.57] | 1.13 [0.89 to 1.44]
  GSK1268997 | 1.02 [0.73 to 1.45] | 0.31 [0.22 to 0.44] | 1.65 [1.19 to 2.27] | 0.84 [0.56 to 1.24]
  GSK1071306 | 0.39 [0.29 to 0.51] | 0.22 [0.16 to 0.29] | 0.61 [0.43 to 0.86] | 0.42 [0.3 to 0.59]

7. Secondary Outcome: Tmax for the Indicated Metabolites of Pazopanib When Administered Alone or in Combination With Ketoconazole and Ezomeprazole
Description: as for outcome 3
Time Frame: as for outcome 1
Population: PK Population
Measure: Median (Full Range); unit: hr
Arm/Group | Pazopanib 400 mg QD | Pazopanib 400 mg QD + Ketoconazole 400 mg QD | Pazopanib 800 mg QD | Pazopanib 800 mg QD + Esomeprazole 40 mg QD
Number analyzed (Participants) | 21 | 16 | 12 | 12
hr
  GSK1268992 | 4 [2 to 24.3] | 24 [0 to 27] | 3 [1.1 to 5.8] | 3 [1 to 24.8]
  GSK1268997 | 3.02 [2 to 8] | 13.4 [0 to 27] | 2.2 [1.1 to 6.1] | 2.4 [1 to 24.8]
  GSK1071306 | 3.12 [2 to 8.9] | 24.1 [0 to 27] | 3.9 [2 to 7.9] | 6 [1 to 24.8]

8. Secondary Outcome: Plasma Ketoconazole Concentration at the Indicated Time Points
Description: Blood samples for the determination of plasma ketoconazole concentrations were collected before (pre-dose [within 60 minutes prior to pazopanib administration]) and after the final pazopanib and ketoconazole dose (fifth dose) during Period 2 at the indicated time points, relative to pazopanib administration (at 1 and 2 hours after pazopanib administration). Blood samples were obtained via peripheral intravenous cannula or central line. Concentrations of ketoconazole were determined in plasma samples using the currently approved analytical methodology.
Time Frame: Day 5 of Period 2 (combination therapy). Blood samples were collected within 60 minutes prior to pazopanib administration and 1 and 2 hours after pazopanib administration.
Population: PK Population
Measure: Mean (Full Range); unit: mcg/mL
Groups:
- Pazopanib 400 mg QD + Ketoconazole 400 mg QD: Pazopanib 400 milligrams (mg) (2x200 mg tablets) once daily (QD), for at least 7 consecutive days in the morning during Period 1, followed by ketoconazole 400 mg (2x200 mg tablets) QD in combination with pazopanib 400 mg (2x200 mg tablets) QD for 5 consecutive days in the morning during Period 2
Arm/Group | Pazopanib 400 mg QD + Ketoconazole 400 mg QD
Number analyzed (Participants) | 16
mcg/mL
  Pre-dose | 0.53 [0 to 1.56]
  1 hr | 4.21 [0.18 to 10.5]
  2 hr | 4.82 [0.24 to 8.40]

9. Secondary Outcome: Number of Participants With the Indicated Grade 3 or 4 Adverse Events (AEs)
Description: AEs were graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 4.0. Grades range from 0 (no toxicity) to 4 (life-threatening or disabling). A Grade 3 AE is severe; defined as considerable interference with the participant's daily activities, medical intervention/therapy required, and hospitalization possible. A Grade 4 AE is life-threatening; defined as extreme limitation in activity, significant medical intervention/therapy required, and hospitalization probable.
Time Frame: From Baseline (Day 1) to a maximum of 4 weeks after the last dose of study drug was administered (on Study Day 12)
Population: All Treated Population: all participants who were enrolled into the study and received at least one dose of study drug
Measure: Number; unit: participants
Arm/Group | Pazopanib 400 mg QD | Pazopanib 400 mg QD + Ketoconazole 400 mg QD | Pazopanib 800 mg QD | Pazopanib 800 mg QD + Esomeprazole 40 mg QD
Number analyzed (Participants) | 21 | 21 | 13 | 13
participants
  Hypertension | 1 | 2 | 0 | 2
  Hypokalemia | 0 | 1 | 0 | 0
  Hypophosphatemia | 0 | 1 | 0 | 0
  Lymphopenia | 0 | 1 | 0 | 0

10. Secondary Outcome: Number of Participants With the Indicated Event of Dose Limiting Toxicity (DLT)
Description: The following were considered DLTs only while participants were receiving pazopanib co-administered with either ketoconazole or esomeprazole: Grade 4 hematologic toxicities, excluding lymphopenia; and Grade 3/4 non-hematologic toxicities, excluding alopecia and nausea/vomiting/diarrhea for which adequate supportive therapy had not been instituted. Toxicities observed once co-administration of pazopanib with ketoconazole or esomeprazole was complete (after Day 5 of Period 2) could also be considered DLTs if judged to be relevant by the investigator and the GlaxoSmithKline Medical Monitor.
Time Frame: From Baseline (Day 1) to a maximum of 4 weeks after the last dose of study drug was administered (on Study Day 12)
Population: All Treated Population. Per protocol, a DLT could not occur during single-agent pazopanib administration in Period 1; thus, data were only collected and analyzed for those participants receiving pazopanib co-administered with either ketoconazole or esomeprazole in Period 2.
Measure: Number; unit: participants
Arm/Group | Pazopanib 400 mg QD | Pazopanib 400 mg QD + Ketoconazole 400 mg QD | Pazopanib 800 mg QD | Pazopanib 800 mg QD + Esomeprazole 40 mg QD
Number analyzed (Participants) | 0 | 21 | 0 | 13
participants |  | 2 |  | 0

ADVERSE EVENTS:
Arm/Group | Pazopanib 400 mg QD | Pazopanib 400 mg QD + Ketoconazole 400 mg QD | Pazopanib 800 mg QD | Pazopanib 800 mg QD + Esomeprazole 40 mg QD
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 11/21 | 17/21 | 2/13 | 8/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib 400 mg QD (N=21) | Pazopanib 400 mg QD + Ketoconazole 400 mg QD (N=21) | Pazopanib 800 mg QD (N=13) | Pazopanib 800 mg QD + Esomeprazole 40 mg QD (N=13)
Nausea (Gastrointestinal disorders) | 5 | 2 | 1 | 2
Vomiting (Gastrointestinal disorders) | 3 | 4 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 2 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oral Discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 4 | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 5 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 4 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1
Blood Bilirubin Increased (Investigations) | 1 | 2 | 0 | 0
Blood Creatinine Increased (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0
Blood Amylase Increased (Investigations) | 0 | 2 | 0 | 0
Activated Partial Thromboplastin Time Prolonged (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 1 | 0 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 1 | 0 | 0
Lipase Increased (Investigations) | 0 | 1 | 0 | 0
White Blood Cell Count Decreased (Investigations) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 3 | 3 | 0 | 3
Asthenia (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 2
Hunger (General disorders) | 1 | 0 | 0 | 0
Mucosal Inflammation (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Gait Disturbance (General disorders) | 0 | 0 | 0 | 1
Edema (General disorders) | 0 | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Adrenal Insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 2 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.